CLINICAL TRIAL: NCT06323499
Title: Outcome After Ablation of Atypical Atrial Flutter: is Induction a Feasible Approach?
Brief Title: Outcome of Induced Atypical Atrial Flutter
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Sponsor
Other Study IDs: UK Essen
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Tachyarrhythmia; Atypical Atrial Flutter; Induction of Arryhthmia; Clinical Outcome
MeSH Terms: conditions — Tachycardia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Induced atypical atrial flutter: Sinus rhythm when starting the procedure, so atypical atrial flutter had to be induced.
  Interventions: Procedure: Induction of atypical atrial flutter
- Ongoing atrial flutter: Atypical atrial flutter was already ongoing when starting the procedure.

INTERVENTIONS:
Procedure: Induction of atypical atrial flutter — Electrophysiological study with induction of atypical atrial flutter. When the induction was successful, ablation of arrhythmia was performed similar to the control group.
  Groups: Induced atypical atrial flutter

SUMMARY:
Background: Atypical atrial flutter (AAF) is an increasingly relevant clinical problem. Despite advancements in mapping and ablation techniques, the general management of these patients remain challenging especially when mapping cannot be performed during ongoing arrhythmia. There are no data whether induction of AAF is a feasible approach in these cases.

Methods: The investigators retrospectively analyzed patients who underwent catheter ablation of AAF and compared procedural results between patients with ongoing tachycardia when starting the procedure and patients with induced AAF.

For this retrospective study, the investigators analyzed patients undergoing ablation of AAF between April 2018 and January 2021 that were identified from the ablation database at the West German Heart and Vascular Center, Essen. All patients were followed up in the outpatient clinic as part of the clinical standard routine or contacted by telephone to assess the occurrence of clinical recurrence of any arrhythmia. In case the documentation was not performed at the institution, relevant documents and ECGs were requested and reviewed.

This single-center cohort study was conducted at the University Hospital Essen, Germany, in accordance with the Declaration of Helsinki and its amendments and was approved by the institutional review board of the University of Essen (number 21-10341-BO). Written informed consent was obtained from all study participants.

The primary study endpoint was to evaluate the outcome of patients with induced AAF in comparison to patients with ongoing AAF when starting the procedure. Furthermore, the investigators analyzed the type of recurrence during follow-up as well as the occurrence and results of repeat ablations at the institution. The investigators also evaluated if the recurrent AAF form was the same or de-novo compared to the AAF during previous procedure.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* symptomatic atypical atrial flutter and electrophysiological study with ablation

Exclusion Criteria:

* inability to comply with follow up
* participation in another trial that may interfere

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic, documented atypical atrial flutter undergoing ablation.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Outcome of patients with induced AAF in comparison to patients with ongoing AAF when starting the procedure. | April 2018 - October 2021
  Recurrence rate of atrial arrhythmias following induced Atrial Fibrillation (AAF) ablation compared to ongoing AAF. The primary outcome measure involves performing ECGs to ascertain the rhythm. When an atrial arrhythmia is confirmed, the patient is categorized as having recurrent arrhythmia. The recurrence rate is calculated as the proportion of cases with documented arrhythmia out of all cases.

SECONDARY OUTCOMES:
Type of recurrence during follow-up | April 2018 - October 2021
  Type of arrhythmia in follow-up: atrial fibrillation, atypical atrial flutter or both. ECGs will be used to determine the type of arrhythmia.
Occurrence and results of repeat ablations at our institution | April 2018 - October 2021
  If patients were re-ablated at the institution, the investigators also evaluated if the recurrent AAF form was the same or de-novo compared to the AAF during previous procedure. Electrophysiological characteristics during procedure are used to determine the form of arrhythmia.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Essen, Essen, North Rhine-Westphalia, Germany